CLINICAL TRIAL: NCT00957021
Title: A Prospective, Post-market, Multi-center Study of the Outcomes of the Triathlon® Posteriorly Stabilized (PS) Total Knee System
Brief Title: Triathlon® Posteriorly Stabilized (PS) Total Knee System - Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon® PS Total Knee System (Other): Triathlon® PS Total Knee System
  Interventions: Device: Triathlon® PS Total Knee System

INTERVENTIONS:
Device: Triathlon® PS Total Knee System — Triathlon® PS Total Knee system

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes (range of motion, pain, function, radiographic stability, and health related quality of life) of patients receiving the Triathlon® Posterior Stabilized (PS) Total Knee System. These outcomes will be evaluated using pre-operative scores and comparing them to post-operative scores in addition to being compared with cases who received the Scorpio® PS implant.

DETAILED DESCRIPTION:
The Triathlon® Posteriorly Stabilized (PS) Total Knee System components are for use in cemented total knee arthroplasty for painful, disabling joint disease of the knee resulting from non-inflammatory degenerative joint disease (including osteoarthritis, traumatic arthritis or avascular necrosis) or rheumatoid arthritis (excluded from this study according to protocol).

The components are designed to improve range of motion (ROM) and stability. This study serves to demonstrate that subjects have reduced pain, increased ROM and improved stability following implantation with the Triathlon® PS Total Knee System.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or non-pregnant female 21-80 years of age at the time of enrollment.
2. The subject requires a primary cemented total knee replacement.
3. The subject has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
4. The subject has intact collateral ligaments.
5. The subject has signed the IRB approved, study specific Informed Patient Consent Form.
6. The subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. The subject has inflammatory arthritis.
2. The subject is morbidly obese, BMI > 40.
3. The subject has a history of total or unicompartmental reconstruction of the affected joint.
4. The subject has had a high tibial osteotomy or femoral osteotomy.
5. The subject has a neuromuscular or neurosensory deficiency that would limit the ability to assess the performance of the device.
6. The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
7. The subject is immunologically suppressed, or receiving chronic steroids (>30 days duration).
8. The subject's bone stock is compromised by disease or infection and cannot provide adequate support and/or fixation to the prosthesis.
9. The subject has had a knee fusion at the affected joint.
10. The subject has an active or suspected latent infection in or about the knee joint.
11. The subject is a prisoner.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2005-12; Primary Completion 2011-03 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Benson, MD, Principal Investigator — New Hampshire Orthopaedic Surgery, PA; Daniel Moretta, DO, Principal Investigator — Tri County Orthopedics Surgeons, Inc.; James Bono, MD, Principal Investigator — New England Baptist Hospital; David W Edelstein, MD, Principal Investigator — Kelsey-Seybold Clinic; Philip Ireland, MD, Principal Investigator — Ireland Hip and Knee Surgery; Joseph P Nessler, MD, Principal Investigator — St. Cloud Orthopaedic Associates; Quanjun Cui, MD, Principal Investigator — University of Virginia; Arnold Scheller, MD, Principal Investigator — Pro-Sports Orthopaedics, Inc./ New England Baptist Hospital; Joel Sorger, MD, Principal Investigator — Wellington Orthopaedics and Sports Medicine; Suresh Nayak, MD, Principal Investigator — Wellington Orthopaedics and Sports Medicine; John I Waldrop, MD, Principal Investigator — Hughston Clinic, PA; James McGrory, MD, Principal Investigator — Hughston Clinic, PA; Steven B Zelicof, MD, PhD, Principal Investigator — Specialty Orthopaedics
Locations (11):
- United States (11):
  - Hughston Clinic PA, Columbus, Georgia
  - Ireland Hip and Knee Surgery, Indianapolis, Indiana
  - New England Baptist Hospital, Boston, Massachusetts
  - Pro-Sports Orthopaedics, Inc. / New England Baptist Hospital, Boston, Massachusetts
  - St. Cloud Orthopaedic Associates, Sartell, Minnesota
  - New Hampshire Orthopaedic Surgery, PA, Manchester, New Hampshire
  - Specialty Orthopaedics, Harrison, New York
  - Wellington Orthopaedics & Sports Medicine, Cincinnati, Ohio
  - Tri County Orthopedic Surgeons, Inc., Massillon, Ohio
  - Kelsey-Seybold Clinic, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 409 participants/500 knees enrolled - 55 participants/65 knees censored = 354 participants/435 knees followed.
Groups:
- Triathlon® PS Total Knee System: If both knees were replaced, but only one knee completed the study, the participant is counted as completed.
Period: Overall Study
Arm/Group | Triathlon® PS Total Knee System
Started | 354
Completed | 237 (Completed/Not completed counts are based on participant status at the 2 yr primary outcome interval.)
Not Completed | 117
Not completed — Death | 5
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 34
Not completed — No 2 yr ROM data | 35
Not completed — Revised study component by 2 yr visit | 8
Not completed — Site Termination by the 2 yr visit | 16
Not completed — Surgery Cancelled | 9
Not completed — Termination due to language issue | 2

BASELINE CHARACTERISTICS:
Population: Participants who were censored protocol violations or who were enrolled, but did not have surgery and age data was not available, are not included in the baseline analysis.
Groups:
- Triathlon® PS Total Knee System: Participants who were not censored from analysis.
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 351
Age, Continuous [Mean (Standard Deviation); unit: years] — For bilateral total knee replacement participants, the age at the time of the initial knee replacement surgery is used.
  3 participants did not have demographic data which would allow calculation of age; these participants did not receive the Triathlon® PS Total Knee System and are part of the "surgery cancelled" participant flow category.
  years | 65.12 (8.59)
Gender [Count of Participants; unit: Participants]
  Female | 200
  Male | 151
Region of Enrollment [Number; unit: participants]
  United States | 351

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion
Description: The primary outcome of this study is to compare active range of motion values for the Triathlon PS Total Knee System.
Time Frame: 2 years
Population: Participants can have both knees replaced. Range of motion is measured for each knee, as such the number of knees evaluated can be greater than the number of participants.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Knees
Groups:
- Triathlon® PS Total Knee System: Includes participants who received the Triathlon® PS Total Knee System. Participants may have bilateral Triathlon® PS Total Knee replacement (TKR), with surgery occurring on different dates. Participants can therefore have a different status for each knee. If one knee has completed the study (i.e. has 2 year ROM data), the participant is counted in the study complete category.
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 237
Number analyzed (Knees) | 291
degrees | 124 (9.98)

2. Secondary Outcome: Patient Outcome Knee Society Score
Description: The Knee Society Scores (KSS) at 1, 2, and 5-year visits will be compared. Additionally, comparison of scores at each post-surgery visit with baseline will be tested to see if any improvement is seen at each time point. The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, ROM and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: 1,2 and 5 years
Population: Maximum number of knees evaluated at any interval.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Groups:
- Triathlon® PS Total Knee System: Includes non-censored participants/knees who received the Triathlon PS Total Knee System. Secondary Objectives are reported by knee.
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 275
Number analyzed (knees) | 340
units on a scale
  Pain/Motion 1 Yr (N=335) | 93.77 (9.03)
  Pain/Motion 1 Yr difference from Baseline (N=333) | 57.36 (16.80)
  Function 1 Yr (N=340) | 86.26 (15.50)
  Function 1 Yr difference from Baseline (N=340) | 30.99 (17.43)
  Pain/Motion 2 Yr (N=281) | 93.96 (8.45)
  Pain/Motion 2 Yr difference from Baseline (N=279) | 57.76 (17.20)
  Function 2 Yr (N=284) | 87.38 (16.40)
  Function 2 Yr difference from Baseline (N=284) | 32.55 (18.89)
  Pain/Motion 5 Yr (N=230) | 94.61 (7.62)
  Pain/Motion 5 Yr difference from Baseline (N=229) | 58.56 (16.35)
  Function 5 Yr (N=232) | 82.07 (20.74)
  Function 5 Yr difference from Baseline (N=232) | 27.33 (22.59)
Statistical Analysis 1: Comparison: Triathlon® PS Total Knee System; KSS Pain/Motion and Function Score comparison from pre-op to 1, 2 and 5 year; Test type: Superiority or Other; p < .0001, t-test, 2 sided

3. Secondary Outcome: Patient Outcome SF-36
Description: The SF-36 score at 1, 2, 3, 4 and 5-year visits will be compared at each post-surgery visit with baseline to see if any improvement is seen for each time point.The SF-36 includes a physical component and a mental component and is completed by the participant. Physical component and mental component scores were calculated on a scale ranging from 0 to 100. Low values represented a poor health state and high values represented a good health state.
Time Frame: 1,2,3,4 and 5 years
Population: Maximum number of knees evaluated at any interval.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 273
Number analyzed (knees) | 335
units on a scale
  SF36 Physical Component 1 Yr (N=335) | 48.16 (8.50)
  SF36 Physical 1 Yr difference from Baseline(N=332) | 15.32 (9.28)
  SF36 Mental Component 1 Yr (N=335) | 55.21 (8.02)
  SF36 Mental 1Yr difference from Baseline(N=332) | 2.58 (11.06)
  SF36 Physical Component 2Yr (N=290) | 47.34 (9.57)
  SF36 Physical 2 Yr difference from Baseline(N=288) | 14.54 (9.75)
  SF36 Mental Component 2 Yr (N=290) | 55.04 (8.10)
  SF36 Mental 2Yr difference from Baseline(N=288) | 2.04 (10.90)
  SF36 Physical Component 3Yr (N=259) | 47.23 (9.31)
  SF36 Physical 3 Yr difference from Baseline(N=257) | 14.45 (9.58)
  SF36 Mental Component 3 Yr (N=259) | 54.30 (9.68)
  SF36 Mental 3 Yr difference from Baseline(N=257) | 1.93 (11.06)
  SF36 Physical Component 4 Yr (N=254) | 46.26 (10.05)
  SF36 Physical 4 Yr difference from Baseline(N=253) | 13.58 (10.54)
  SF36 Mental Component 4 Yr (N=254) | 54.49 (8.74)
  SF36 Mental 4 Yr difference from Baseline(N=253) | 1.93 (10.88)
  SF36 Physical Component 5 Yr (N=243) | 46.33 (9.72)
  SF36 Physical 5 Yr difference from Baseline(N=242) | 13.65 (10.82)
  SF36 Mental Component 5 Yr (N=243) | 54.82 (7.97)
  SF36 Mental 5 Yr difference from Baseline(N=242) | 2.25 (11.06)
Statistical Analysis 1: Comparison: Triathlon® PS Total Knee System; SF-36 Physical score comparison from pre-op to 1, 2, 3, 4 and 5 years; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Triathlon® PS Total Knee System; SF-36 Mental score comparison from pre-op to 1 year; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Triathlon® PS Total Knee System; SF-36 Mental score comparison from pre-op to 2 year; Test type: Superiority or Other; p = 0.0017, t-test, 2 sided
Statistical Analysis 4: Comparison: Triathlon® PS Total Knee System; SF-36 Mental score comparison from pre-op to 3 year; Test type: Superiority or Other; p = 0.0055, t-test, 2 sided
Statistical Analysis 5: Comparison: Triathlon® PS Total Knee System; SF-36 Mental score comparison from pre-op to 4 year; Test type: Superiority or Other; p = 0.0050, t-test, 2 sided
Statistical Analysis 6: Comparison: Triathlon® PS Total Knee System; SF-36 Mental score comparison from pre-op to 5 year; Test type: Superiority or Other; p = 0.0018, t-test, 2 sided

4. Secondary Outcome: Patient Outcome WOMAC
Description: The Western Ontario and McMaster Osteoarthritis Index (WOMAC) scores at 1, 2, 3, 4 and 5-year visits will be compared between groups, when data is available. Additionally, comparison of scores at each post-surgery visit with baseline will be tested to see if any improvement is seen for each time point. The WOMAC collects information specific to osteoarthritis outcomes. The questionnaire uses a visual analog scale for pain, measuring factors of general pain, stiffness, and physical findings. Pain is scored from 0 to 100 for each set of factors, with 0 indicating no pain and 100 indicating extreme pain. Total WOMAC scores range from 0 to 300. Lower values represent better outcomes.
  Data for the WOMAC is only available at the 5 year interval due to typographical errors noted on earlier interval forms rendering them invalid for comparison.
Time Frame: 5 years
Population: The number of knees evaluated at 5 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 197
Number analyzed (knees) | 236
units on a scale | 45.11 (53.96)

5. Secondary Outcome: Patient Outcome Lower-Extremity Activity Scale
Description: The Lower-Extremity Activity Scale (LEAS) score at 1, 2, 3, 4 and 5-year intervals will be compared at each post-surgery visit with baseline to see if any improvement is seen for each time point.The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level. A level of 1 indicated that the subject was confined to bed all day while a level of 18 indicated that the subject was up and about at will inside and outside of the house, and also participated in vigorous physical activity, such as competitive level sports, on a daily basis.
Time Frame: 1,2,3,4 and 5 years
Population: Maximum number of knees available at any interval.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 274
Number analyzed (knees) | 339
units on a scale
  LEAS 1 Year (N=339) | 11.22 (2.62)
  LEAS 1 Year difference from Baseline (N=339) | 1.97 (2.84)
  LEAS 2 Year (N=291) | 11.04 (2.63)
  LEAS 2 Year difference from Baseline (N=291) | 1.86 (2.98)
  LEAS 3 Year (N=266) | 11.15 (2.87)
  LEAS 3 Year difference from Baseline (N=266) | 1.95 (3.12)
  LEAS 4 Year (N=262) | 10.97 (2.76)
  LEAS 4 Year difference from Baseline (N=262) | 1.87 (3.03)
  LEAS 5 Year (N=244) | 11.02 (2.93)
  LEAS 5 Year difference from Baseline (N=244) | 1.89 (3.14)
Statistical Analysis 1: Comparison: Triathlon® PS Total Knee System; LEAS score comparison from pre-op to 1, 2, 3, 4 and 5 years; Test type: Superiority or Other; p < .0001, t-test, 2 sided

6. Secondary Outcome: Radiographic Outcome
Description: Radiographic success/failure at 1, 2, and 5-year visits will be assessed. Radiographic failure is defined as a score of 10 or greater according to the Knee Society Roentgenographic Scoring System, regardless of symptoms. A migrating or shifting prosthesis with or without the disappearance of radiolucent lines is also a failure regardless of score.
Time Frame: 1,2 and 5 years
Population: Maximum number of knees evaluable at any interval.
Measure: Number; unit: knees
Units Other Than Participants: knees
Arm/Group | Triathlon® PS Total Knee System
Number analyzed (Participants) | 311
Number analyzed (knees) | 345
knees
  Radiographic failure at 1 Yr (N=347 knees) | 1
  Radiographic failure at 2 Yrs (N=282 knees) | 2
  Radiographic failure at 5 Yrs (N=217 knees) | 3

ADVERSE EVENTS:
Time Frame: This study requires that all operative site and systemic adverse events be reported from enrollment to 5 years postoperative. This includes any change from baseline status. Censored protocol violations were not included as at risk participants.
Description: Elective procedures are not included. These may include: non-study total knee/hip replacements/revisions, rotator cuff repairs, carpal tunnel releases, cataract & intra-ocular procedures, bunion procedures, total shoulder repairs, laminectomies, microdiscectomies, breast reductions, cervical spine fusions, & mid-foot/flat-foot surgeries.
Groups:
- Triathlon® PS Total Knee System: All non-censored participants who received the Triathlon® PS Total Knee System.
Arm/Group | Triathlon® PS Total Knee System
Serious Adverse Events (participants affected / at risk) | 86/354
Other Adverse Events (participants affected / at risk) | 194/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon® PS Total Knee System (N=354)
Non-operative site (Cardiac disorders) | 15 (17)
Non-operative site (Gastrointestinal disorders) | 9 (10)
Non-operative Site (General disorders) | 2 (3)
Non-operative Site (Immune system disorders) | 1 (1)
Operative Site (Infections and infestations) | 8 (8)
Non-operative Site (Infections and infestations) | 3 (3)
Operative Site (Injury, poisoning and procedural complications) | 2 (2)
Non-operative Site (Metabolism and nutrition disorders) | 1 (1)
Operative Site (Musculoskeletal and connective tissue disorders) | 21 (22)
Non-operative Site (Musculoskeletal and connective tissue disorders) | 16 (19)
Non-operative Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Non-operative Site (Nervous system disorders) | 4 (4)
Non-operative Site (Psychiatric disorders) | 1 (1)
Non-operative Site (Renal and urinary disorders) | 3 (3)
Non-operative Site (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Non-operative Site (Vascular disorders) | 3 (4)
Operative Site (Nervous system disorders) | 1 (1)
Non-operative Site (Ear and labyrinth disorders) | 1 (1)
Non-operative Site (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon® PS Total Knee System (N=354)
Operative Site (Musculoskeletal and connective tissue disorders) | 90 (121)
Non-operative Site (Musculoskeletal and connective tissue disorders) | 111 (203)
Non-operative Site (Respiratory, thoracic and mediastinal disorders) | 29 (65)
Non-operative Site (Blood and lymphatic system disorders) | 31 (34)
Non-operative Site (Gastrointestinal disorders) | 27 (34)
Non-operative Site (Nervous system disorders) | 24 (29)
Non-operative Site (Renal and urinary disorders) | 22 (30)
Non-operative Site (Skin and subcutaneous tissue disorders) | 26 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study. These manuscripts and abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.